CLINICAL TRIAL: NCT05574556
Title: Electromiographic Analysis of the Quadriceps in Individuals Undergoing Neuromuscular Electro-stimulation Intervention, Verbal Command and Neuromatrix
Brief Title: Electromiographic Analysis of the Quadriceps After Trauma
Status: Completed | Type: Observational
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: Electromiographic Analysis
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Leg Injury; Bone Fracture
MeSH Terms: conditions — Leg Injuries; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- myoelectric activity of the quadriceps muscle: electromyography myoelectric activity of the quadriceps muscle

SUMMARY:
The lower limb is the region most affected by fractures in the human body. The magnitude of the trauma can cause injuries to structures adjacent to the fracture, promoting joint instability and consequently predisposition to osteoarthritis. The treatment of fractures can be performed conservatively or surgically, and one of the consequences of the surgery is arthrogenic muscle inhibition, which presents itself as a marked muscle weakness due to inhibition of the central nervous system that prevents adequate muscle activation. However, recruiting the quadriceps is the most commonly used goal to determine the patient's return to activities. Physiotherapy has several resources for the functional activation of the quadriceps muscle, such as neuromuscular electrostimulation (NMES), verbal command of muscle activation and neuromatrix techniques. Thus, the objective of this study will be to analyze, by means of electromyography, the myoelectric activity of the quadriceps muscle in individuals undergoing physical therapy intervention, affected by some fracture of the lower limb.

ELIGIBILITY:
Inclusion Criteria:

* trauma in lower member intervention

Exclusion Criteria:

* neuromuscular disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: ANALYSIS OF THE QUADRICEPS AFTER TRAUMA IN LOWER MEMBERSINTERVENTION
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
electromyography | one time - during the procedure
  will be performed an examination of electrical muscle conductance

SECONDARY OUTCOMES:
myoelectric activity of the quadriceps muscle | one time - during the procedure
  will be performed an examination of electrical muscle conductance

CONTACTS AND LOCATIONS:
Locations (1):
- Claudio Cazarini Júnior, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No